CLINICAL TRIAL: NCT04750824
Title: Assessment of Real-World Outcomes Associated With Afatinib (Gilotrif) Use in Patients With Solid Tumors Harboring NRG1 Gene Fusions
Brief Title: Real-World Effectiveness of Afatinib (Gilotrif) Following Immunotherapy in the Treatment of Metastatic, Squamous Cell Carcinoma of the Lung: A Multi-Site Retrospective Chart Review Study in the U.S.
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1200-0335
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Non-squamous, Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- All afatinib patients
  Interventions: Drug: Afatinib
- All non-afatinib (other systemic therapies)
  Interventions: Drug: other systemic therapy

INTERVENTIONS:
Drug: Afatinib — Afatinib
  Other Names: Gilotrif®
  Groups: All afatinib patients
Drug: other systemic therapy — other systemic therapy
  Groups: All non-afatinib (other systemic therapies)

SUMMARY:
Characteristics of patients with Neuregulin-1 (NRG1) gene fusion-positive solid tumors treated with afatinib, and characteristics of those treated with another systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 years of age or older, at the time of diagnosis with any solid tumor.
* Confirmed NRG1 gene fusion in any solid tumor.
* Initiated afatinib or other systemic therapy (in any line of therapy) for treatment of a solid tumor with NRG1 gene fusion on or after 01/01/2017 through 03/31/2020.
* Followed up for ≥3 months after initiation of afatinib or other systemic therapy (unless deceased prior to 3 months of follow-up).

Exclusion Criteria:

- Treatment with any Tyrosine kinase inhibitor (TKI)/ErbB-directed therapy other than afatinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Providers will select patients meeting the study eligibility criteria as described below. Providers will be asked to select eligible patients chronologically, starting with the first patient who first initiated any line of afatinib or chemotherapy, on or after 01/01/2017 through 03/31/2020.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cardinal Health, Dublin, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-interventional, retrospective, United States (US), multi-site, cohort study based on existing data from medical records of patients with Neuregulin-1 (NRG1) gene fusion-positive solid tumors treated with afatinib or other systemic therapy.
Pre-assignment Details: Only subjects that met all inclusion and none of the exclusion criteria were included.
Groups:
- All Afatinib Patients: Patients with a confirmed Neuregulin-1 (NRG1) gene fusion in any solid tumor, who initiated treatment with afatinib (in any line of therapy) for treatment of a solid tumor with NRG1 gene fusion on or after 01-January-2017 through 31-March-2020 and followed up for ≥3 months after initiation of afatinib (unless deceased prior to 3 months of follow-up).
- All Non-afatinib (Other Systemic Therapies): Patients with a confirmed Neuregulin-1 (NRG1) gene fusion in any solid tumor, who initiated treatment with other systemic therapies than afatinib (in any line of therapy) for treatment of a solid tumor with NRG1 gene fusion on or after 01-January-2017 through 31-March-2020 and followed up for ≥3 months after initiation of other systemic therapies than afatinib (unless deceased prior to 3 months of follow-up).
Period: Overall Study
Arm/Group | All Afatinib Patients | All Non-afatinib (Other Systemic Therapies)
Started | 72 | 38
First Line Therapy Patients | 16 | 36
Completed (Patients receiving index therapy at data collection (i.e.11-November-2020 to 20-January-2021)) | 10 | 14
Not Completed | 62 | 24
Not completed — Toxicity/intolerability | 3 | 1
Not completed — Death | 1 | 3
Not completed — Scheduled duration of therapy complete | 1 | 9
Not completed — Disease progression (confirmed with scan) | 57 | 11

BASELINE CHARACTERISTICS:
Population: All patients who initiated index therapy (i.e., afatinib in any line; other systemic therapy among those without any history of afatinib) between 01 January 2017 and 31 March 2020.
Groups:
- Total: Total of all reporting groups
Arm/Group | All Afatinib Patients | All Non-afatinib (Other Systemic Therapies) | Total
Number analyzed (Participants) | 72 | 38 | 110
Age, Continuous [Median (Inter-Quartile Range); unit: Years] — Age at initiation of index therapy.
  Years | 62 [58 to 68] | 66 [59 to 71] | 62.5 [59.0 to 70.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 18 | 48
  Male | 42 | 20 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 5 | 15
  Not Hispanic or Latino | 62 | 33 | 95
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 16 | 16 | 32
  White | 48 | 22 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Geographic Region [Count of Participants; unit: Participants] — Number of patients in each category of Geographic Region is reported. The reported categories of geographic region are:
  Northeast; Midwest; South; West.
  Participants
    Northeast | 26 | 10 | 36
    Midwest | 5 | 4 | 9
    South | 15 | 24 | 39
    West | 26 | 0 | 26
Line of therapy in which index therapy was received [Count of Participants; unit: Participants] — Number of patients in each category of line of therapy in which index therapy was received is reported.
  The reported categories of line of therapy are:
  First line (1L); Second line (2L);
  * third line (3L+).
  Participants
    First line therapy (1L) | 16 | 36 | 52
    Second line therapy (2L) | 51 | 2 | 53
    ≥ third line therapy (3L+) | 5 | 0 | 5
Eastern Cooperative Oncology Group Performance Status (ECOG-PS) [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group Performance Status (ECOG-PS) describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). It is measured on a 6 point scale, from 0 to 5, with 0 meaning the patient is fully active without restrictions and 5 death.
  Number of patients in each reported category of ECOG-PS at the time of initiation of index therapy is reported. The reported categories of ECOG-PS are:
  0 or 1; 2+ (i.e.. includes 2,3,4).
  Participants
    0,1 | 22 | 26 | 48
    2+ | 50 | 12 | 62
Smoking status at initiation of index therapy [Count of Participants; unit: Participants] — Number of patients in each category of smoking status at initiation of index therapy. The reported categories of smoking status are:
  Never smoked; Current smoker; Past history of smoking.
  Participants
    Never smoked | 32 | 14 | 46
    Current smoker | 2 | 2 | 4
    Past history of smoking | 38 | 22 | 60
Tumor stage at initiation of index therapy [Count of Participants; unit: Participants] — Number of patients in each category of tumor stage at initiation of index therapy is reported. The reported categories of tumor stage are:
  Stage I; Stage II; Stage III; Stage IV.
  Participants
    Stage I | 0 | 0 | 0
    Stage II | 1 | 3 | 4
    Stage III | 6 | 1 | 7
    Stage IV | 65 | 34 | 99
Comorbidities [Count of Participants; unit: Participants] — Number of patients in each category of comorbidities. The reported categories of comorbidities are:
  Hypertension; Cardiovascular disease; Diabetes with chronic complications; Chronic pulmonary disease; None of the above.
  Participants
    Hypertension | 29 | 21 | 50
    Cardiovascular disease | 0 | 14 | 14
    Diabetes with chronic complications | 0 | 12 | 12
    Chronic pulmonary disease | 16 | 12 | 28
    Depression | 17 | 0 | 17
    None of the above | 15 | 10 | 25
NRG1 testing characteristics: NRG1 testing location [Count of Participants; unit: Participants] — Number of patients in each category of Neuregulin 1 (NRG1) testing locations is reported. The reported categories of NRG1 testing locations are: Caris Life Sciences; Foundation One; Other; Specialty gene testing lab; Tempus; Unknown.
  Participants
    Caris Life Sciences | 15 | 0 | 15
    Foundation One | 29 | 27 | 56
    Other | 3 | 1 | 4
    Specialty gene testing lab | 11 | 7 | 18
    Tempus | 3 | 0 | 3
    Unknown | 11 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR): Based on Charted/Physician-reported Disease Response
Description: ORR was defined as the percentage of patients with a complete response (CR) or partial response (PR) out of all patients (CR+PR/all patients) at initial response assessment and best response (response based on the scan where the patient showed the best response to treatment (not progression)).
  Charted/physician-reported (physician-provided information as recorded in patient's chart) ORR is reported.
Time Frame: From the index date (i.e., anytime between 01-January-2017 and 31-March-2020) until data collection (i.e. 11-Nov-2020 to 20-Jan-2021), up to 4 years and 19 days.
Population: as for baseline characteristics
Measure: Number; unit: percentage of patients
Groups:
- First Line Afatinib Patients: Patients with a confirmed Neuregulin-1 (NRG1) gene fusion in any solid tumor, who initiated treatment with afatinib as a first line (IL) of therapy for treatment of a solid tumor with NRG1 gene fusion on or after 01-January-2017 through 31-March-2020 and followed up for ≥3 months after initiation of afatinib (unless deceased prior to 3 months of follow-up).
- First Line Non-afatinib Patients: Patients with a confirmed Neuregulin-1 (NRG1) gene fusion in any solid tumor, who initiated treatment with other systemic therapies than afatinib as a first line (IL) of therapy for treatment of a solid tumor with NRG1 gene fusion on or after 01-January-2017 through 31-March-2020 and followed up for ≥3 months after initiation of other systemic therapies than afatinib (unless deceased prior to 3 months of follow-up).
Arm/Group | All Afatinib Patients | All Non-afatinib (Other Systemic Therapies) | First Line Afatinib Patients | First Line Non-afatinib Patients
Number analyzed (Participants) | 72 | 38 | 16 | 36
percentage of patients | 37.5 | 76.3 | 43.8 | 77.8

2. Primary Outcome: Objective Response Rate (ORR): Based on Lesion Measurements and RECIST v1.1 Criteria
Description: ORR based on lesion measurements and RECIST v1.1 criteria is reported. ORR was defined as the percentage of patients with a complete response (CR) or partial response (PR) out of all patients (CR+PR/all patients) at initial response assessment and best response.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1):
  CR: Disappearance of all target lesions or disappearance of all non-target lesions.
  PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: percentage of patients
Groups:
- First Line Afatinib Patients: Patients with a confirmed Neuregulin-1 (NRG1) gene fusion in any solid tumor, who initiated treatment with afatinib as a first line (1L) of therapy for treatment of a solid tumor with NRG1 gene fusion on or after 01-January-2017 through 31-March-2020 and followed up for ≥3 months after initiation of afatinib (unless deceased prior to 3 months of follow-up).
Arm/Group | All Afatinib Patients | All Non-afatinib (Other Systemic Therapies) | First Line Afatinib Patients | First Line Non-afatinib Patients
Number analyzed (Participants) | 72 | 38 | 16 | 36
percentage of patients | 34.7 | 71.1 | 43.8 | 72.2

3. Primary Outcome: Duration of Objective Response (DOR)
Description: DOR was defined as the time from initial response (for any patient with a complete or partial response initially) until the earliest of either disease progression or death. Duration of response is reported for those patients who had a complete or partial response according to charted/physician-reported disease response. Patients who discontinued therapy due to a reason other than progression were censored on the date of discontinuation. Patients still on therapy at the time of data cut-off were censored on their last visit date.
Time Frame: as for outcome 1
Population: All patients who initiated index therapy (i.e., afatinib in any line; other systemic therapy among those without any history of afatinib) between 01 January 2017 and 31 March 2020 and had a complete or partial response according to charted/physician-reported disease response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Afatinib Patients | All Non-afatinib (Other Systemic Therapies) | First Line Afatinib Patients | First Line Non-afatinib Patients
Number analyzed (Participants) | 27 | 29 | 7 | 28
months | 5.851 [3.419 to 9.040] | 13.38 [8.974 to 13.38] | NA [NA to NA] — Median and 95% Confidence Interval could not be calculated due to insufficient number of participants with the event | 13.38 [8.98 to 13.38]

4. Primary Outcome: Duration of Clinical Benefit (DOCB)
Description: DOCB was defined as the time from initial response (for any patient with a complete, partial, or stable disease response initially) until the earliest of either disease progression or death. DOCB reported for those patients who had a complete, partial or response according to charted/physician-reported disease response. Patients who discontinued therapy due to a reason other than progression were censored on the date of discontinuation.
  Patients still on therapy at the time of data cut-off were censored on their last visit date.
Time Frame: as for outcome 1
Population: All patients who initiated index therapy (i.e., afatinib in any line; other systemic therapy among those without any history of afatinib) between 01 January 2017 and 31 March 2020 and had a complete, partial, or stable disease response according to charted/physician-reported disease response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Afatinib Patients | All Non-afatinib (Other Systemic Therapies) | First Line Afatinib Patients | First Line Non-afatinib Patients
Number analyzed (Participants) | 35 | 32 | 8 | 31
months | 5.85 [2.99 to 9.04] | 13.38 [8.97 to 13.38] | NA [NA to NA] — Could not be calculated due to insufficient number of participants with events. | 13.38 [8.97 to 13.38]

5. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as time from initiation of a line of therapy until disease progression or death; patients on therapy at the time of data cut-off were censored on the last date of treatment. Patients who discontinued a line of therapy for a reason other than disease progression but who subsequently die prior to the receipt of any other therapy were considered an event on the date of death.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1):
  Progressive disease (PD): at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study), or unequivocal progression of existing non-target lesions, or the appearance of one or more new lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 millimeter (mm).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Afatinib Patients | All Non-afatinib (Other Systemic Therapies) | First Line Afatinib Patients | First Line Non-afatinib Patients
Number analyzed (Participants) | 72 | 38 | 16 | 36
months | 5.490 [4.602 to 5.917] | 12.886 [4.865 to NA] — Upper Limit of 95% Confidence Interval could not be calculated due to insufficient number of participants with the event. | 6.345 [5.325 to NA] — Upper Limit of 95% Confidence Interval could not be calculated due to insufficient number of participants with the event. | 12.89 [4.865 to NA] — Upper Limit of 95% Confidence Interval could not be calculated due to insufficient number of participants with the event.

6. Primary Outcome: Time on Treatment (TOT)
Description: TOT was defined as time from initiation of a line of therapy until discontinuation for any reason. Patients on therapy at the time of data cut-off were censored on the last date of treatment.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Afatinib Patients | All Non-afatinib (Other Systemic Therapies) | First Line Afatinib Patients | First Line Non-afatinib Patients
Number analyzed (Participants) | 72 | 38 | 16 | 36
months | 5.42 [4.24 to 5.82] | 5.08 [3.48 to 15.91] | 6.34 [5.33 to NA] — Upper Limit of 95% Confidence Interval could not be calculated due to insufficient number of participants with the event. | 5.08 [3.48 to 15.91]

7. Primary Outcome: Time to Progression (TTP)
Description: TTP was defined as time from initiation of a line of therapy until discontinuation due to disease progression. Patients on therapy or those who discontinued due to a reason other than disease progression were censored on the last date of treatment.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Groups:
- First Line Non-afatinib Patients: Patients with a confirmed Neuregulin-1 (NRG1) gene fusion in any solid tumor, who initiated treatment with other systemic therapies than afatinib as a first line of therapy for treatment of a solid tumor with NRG1 gene fusion on or after 01-January-2017 through 31-March-2020 and followed up for ≥3 months after initiation of other systemic therapies than afatinib (unless deceased prior to 3 months of follow-up).
Arm/Group | All Afatinib Patients | All Non-afatinib (Other Systemic Therapies) | First Line Afatinib Patients | First Line Non-afatinib Patients
Number analyzed (Participants) | 72 | 38 | 16 | 36
months | 5.49 [4.60 to 6.08] | 12.89 [12.89 to NA] — Upper Limit of 95% Confidence Interval could not be calculated due to insufficient number of participants with the event. | 6.44 [5.36 to NA] — Upper Limit of 95% Confidence Interval could not be calculated due to insufficient number of participants with the event. | 12.89 [12.89 to NA] — Upper Limit of 95% Confidence Interval could not be calculated due to insufficient number of participants with the event.

8. Primary Outcome: Overall Survival (OS)
Description: OS was defined as time from initiation of any therapy in the metastatic setting until death. Patients alive at the time of data cut-off were censored on the last date the patient was seen by the provider/clinic.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Afatinib Patients | All Non-afatinib (Other Systemic Therapies) | First Line Afatinib Patients | First Line Non-afatinib Patients
Number analyzed (Participants) | 72 | 38 | 16 | 36
months | 7.166 [6.246 to 9.040] | 22.551 [10.815 to 29.848] | 9.928 [7.002 to NA] — Upper Limit of 95% Confidence Interval could not be calculated due to insufficient number of participants with the event. | 22.55 [10.82 to 29.85]

9. Primary Outcome: Number of Patients Who Experienced Any ADRs During Index Treatment Line
Description: Number of patients who experienced any averse drug reactions (ADRs) during index treatment line is reported.
  An ADR was defined as a response to a medicinal product which is noxious and unintended. Response in this context means that a causal relationship between a medicinal product and an adverse event (AE) is at least a reasonable possibility.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | All Afatinib Patients | All Non-afatinib (Other Systemic Therapies) | First Line Afatinib Patients | First Line Non-afatinib Patients
Number analyzed (Participants) | 72 | 38 | 16 | 36
Participants | 7 | 8 | 2 | 8

ADVERSE EVENTS:
Time Frame: From the index date (i.e., anytime between 01-January-2017 and 31-March-2020) until data collection (i.e.11-Nov-2020 to 20-Jan-2021), up to 4 years and 19 days.
Description: All patients who initiated index therapy (i.e., afatinib in any line; other systemic therapy among those without any history of afatinib) between 01 January 2017 and 31 March 2020.
Arm/Group | All Afatinib Patients | All Non-afatinib (Other Systemic Therapies)
All-Cause Mortality (participants affected / at risk) | 1/72 | 3/38
Serious Adverse Events (participants affected / at risk) | 0/72 | 4/38
Other Adverse Events (participants affected / at risk) | 2/72 | 3/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Afatinib Patients (N=72) | All Non-afatinib (Other Systemic Therapies) (N=38)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Afatinib Patients (N=72) | All Non-afatinib (Other Systemic Therapies) (N=38)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT04750824/Prot_SAP_000.pdf